CLINICAL TRIAL: NCT03242889
Title: A Phase 1 Study of Subcutaneous Delivery of JNJ-54767414 (Daratumumab) in Japanese Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Subcutaneous Delivery of JNJ-54767414 (Daratumumab) in Japanese Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108337; 54767414MMY1008 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DARA SC (Experimental): Participants will receive DARA SC (daratumumab 1800 milligram [mg] with Recombinant Human Hyaluronidase [rHuPH20] 30,000 units [U] that is 2000 U/milliliter [U/mL]) subcutaneous (SC) injection once weekly for the first 8 weeks in Cycles 1 and 2 (Days 1, 8, 15, and 22 of each week), every 2 weeks in Cycles 3 to 6 (Days 1 and 15) for the following 16 weeks and then every 4 weeks (from Cycle 7 [Day 1]) in subsequent cycles until disease progression, unacceptable toxicity, or any other reason for discontinuation. Each cycle is 28 days in duration.
  Interventions: Drug: DARA SC

INTERVENTIONS:
Drug: DARA SC — Participants will receive 1800 mg daratumumab with 30,000 U (2000 U/mL) rHuPH20 SC injection once weekly for the first 8 weeks in Cycles 1 and 2 and every 2 weeks in Cycles 3 to 6 for 16 weeks and then every 4 weeks in subsequent cycles until disease progression, unacceptable toxicity, or any other reason for discontinuation.

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of subcutaneous (SC) delivery of co-formulated daratumumab and rHuPH20 preparation (DARA SC) in Japanese participants with relapsed or refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Participant proven to have Multiple Myeloma (MM) according to the International Myeloma Working Group (IMWG) diagnostic criteria
* Participant must have measurable, secretory disease as defined by any of the following:

  1. Immunoglobulin (Ig) G MM: serum M-protein level greater than or equal to (>=) 1.0 gram per deciliter (g/dL) or urine M-protein level >= 200 milligram (mg)/24 hours; or
  2. IgA, IgD, IgE MM: serum M-protein level >= 0.5 g/dL or urine M-protein level >= 200 mg/24 hours; or
  3. Light chain MM, for participants without measurable disease in the serum or urine: serum Ig free light chains (FLC) >= 10 mg/dL and abnormal serum Ig kappa lambda FLC ratio
* Participant must have received >= 2 prior lines of antimyeloma therapy without further established treatment option
* Participant must have relapsed or refractory disease
* Participant must have an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* The Participant must meet the following criteria of clinical laboratory test results during screening phase:

  1. hemoglobin >=7.5 g/dL (>=5 millimoles/liter [mmol/L]) (without prior Red Blood Cells (RBC) transfusion within 7 days before the laboratory test;
  2. absolute neutrophil count (ANC) >=1.0*10^9/L (without granulocyte colony stimulating factor support in the 7 days prior the laboratory test);
  3. platelet count >=75*10^9/L for participants in whom less than (<)50.0 percent (%) of bone marrow nucleated cells are plasma cells; otherwise platelet count >=50*10^9/L (without transfusion support in the 7 days prior to the laboratory test);
  4. aspartate aminotransferase (AST) less than or equal to (<=)3.0 times upper limit of normal (ULN);
  5. alanine aminotransferase (ALT) <=3.0 times ULN;
  6. creatinine clearance >20 mL/minute/1.73 m^2;
  7. total bilirubin <=2.0 times ULN, except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin <=1.5 times ULN is required);
  8. corrected serum calcium <=14 mg/dL (<=3.5 mmol/L)
* Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use highly effective methods of reliable birth control. Contraception must begin 4 weeks before initiating treatment, during therapy, during dose interruptions, and continue for 6 months following discontinuation of study therapy
* A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control, even if he had a successful vasectomy, for example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 6 months after receiving the final dose of study drug

Exclusion Criteria:

* Participant has received daratumumab or other anti cluster of differentiation (CD)38 therapies previously
* Participant has received antimyeloma treatment within 2 weeks before Cycle 1 Day 1
* Participant has received autologous stem cell transplantation (ASCT) within 12 weeks before Cycle 1 Day 1, or the participant has previously received an allogenic stem cell transplant (regardless of timing)
* Participant has received a cumulative dose of corticosteroids equivalent or more than the equivalent of 140 mg of prednisolone within the 2-week period before Cycle 1 Day 1
* Participant has a history of malignancy (other than MM) within 3 years before Cycle 1 Day 1 (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix or breast, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events Including Dose Limiting Toxicity | Up to 30 days after last study drug dose (approximately up to 1 year)
  An adverse event (AE) is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Daratumumab | Up to 8 weeks after the last dose of study drug (approximately up to 1 year)
  Maximum observed concentration of daratumumab will be measured.
Maximum Serum Trough Concentration (Ctrough) of Daratumumab | At Cycle 3 Day 1 predose concentration
  Ctrough is the concentration of daratumumab prior to the next drug administration.
Serum Concentration of Daratumumab and Recombinant Human Hyaluronidase (rHuPH20) (Plasma) Antibodies | Up to 8 weeks after the last dose of study drug (approximately up to 1 year)
  Serum levels of antibodies to daratumumab and rHuPH20 will be analyzed for evaluation of potential immunogenicity.
Overall Response Rate | Approximately up to 1 year
  Overall Response is partial response (PR)/better as per International Myeloma Working Group (IMWG) criteria. PR: >=50% reduction of serum M-protein, >=90% reduction in 24 hour urinary M-protein or to <200 mg/24 hours; if serum and urine M-protein are not measurable, >=50% decrease in difference between involved and uninvolved free light chains (FLC) levels; if serum and urine M-protein and serum free light assay is not measurable, >=50% reduction in bone marrow plasma cell (PC), with baseline bone marrow PC percentage >=30%; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; Very good partial response: serum and urine M-component detectable by immunofixation or >=90.0% reduction in serum M-protein and urine M-protein <100mg/24 hours; Complete response (CR):negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5.0% PCs in bone marrow; Stringent complete response (sCR): CR plus normal FLC ratio and absence of clonal PCs.
Duration of Response (DOR) | First documentation of confirmed PR or better to the date of first documented progressive disease (PD), or date of death due to PD, whichever occurs first (approximately up to 1 year)
  DOR is date of first documentation of confirmed PR or better to date of first documented PD (as per IMWG criteria), or date of death due to PD, whichever occurs first. PD: 25% increase from lowest response value in 1 of following: serum M-component, urine M-component (absolute increase must be >= 0.5 gram per deciliter [g/dL], >= 200 mg/24 hours respectively), Only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase must be >10 milligram per deciliter (mg/dL), only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC% (absolute percentage must be >=10%), definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or tissue plasmacytomas and development of hypercalcemia (serum calcium >11.5 mg/dL) attributed solely to PC proliferative disorder.
Time to Response | Approximately up to 1 year
  Time to response is defined as the time between Cycle 1 Day 1 and the first efficacy evaluation date that the participant has met all criteria for PR or better (as per IMWG criteria). PR: >=50% reduction of serum M-protein, >=90% reduction in 24 hour urinary M-protein or to <200 mg/24 hours; if serum and urine M-protein are not measurable, >=50% decrease in difference between involved and uninvolved FLC levels; if serum and urine M-protein and serum free light assay is not measurable, >=50% reduction in bone marrow PC, with baseline bone marrow PC percentage >=30%; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; Very good partial response: serum and urine M-component detectable by immunofixation or >=90.0% reduction in serum M-protein and urine M-protein <100mg/24 hours; CR: negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5.0% PCs in bone marrow; sCR: CR plus normal FLC ratio and absence of clonal PCs.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (5):
- Japan (5):
  - National Hospital Organization Shibukawa Medical Center, Gunma
  - Nagoya City University Hospital, Nagoya
  - Ogaki Municipal Hospital, Ohgaki
  - Osaka University Hospital, Osaka
  - Japanese Red Cross Medical Center, Shibuya City

REFERENCES:
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- [Derived] Shibayama H, Matsumoto M, Kosugi H, Shibayama K, Yamazaki H, Iida S. Subcutaneous delivery of daratumumab in Japanese patients with relapsed/refractory multiple myeloma. Int J Hematol. 2021 Jan;113(1):112-121. doi: 10.1007/s12185-020-02985-9. Epub 2020 Sep 11. PMID 32915384